CLINICAL TRIAL: NCT03610958
Title: Prospective, Single Center, Open-labeled Single Arm Study, to Asses the Safety and Performance Evaluation of the Epitomee Device for Enhancing Satiety and Weight Loss in Healthy Over Weight and Obese Subjects
Brief Title: Safety and Performance Evaluation of the Epitomee Device for Enhancing Satiety and Weight Loss.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Epitomee medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRT-05-022
Record Dates: First submitted 2018-07-09; First posted 2018-08-01 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Overweight; Obesity
Keywords: overweight; obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Prospective, single center, open-labeled single arm study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epitomee Device arm (Experimental): A non-surgical, non-pharmacologic, medical Device designed to enhance the feeling of satiety. The Device is composed of a 000 size standard capsule and the Tulip's proprietary Device, encapsulated within it.
  The Device components are produced from approved pharmaceutical excipients / food additives / generally recognized as safe (GRAS )/ food contact materials which are used at high grade
  Interventions: Device: Epitomee Device

INTERVENTIONS:
Device: Epitomee Device — A non-surgical, non-pharmacologic, medical Device designed to enhance the feeling of satiety.
  Other Names: Tulip Device

SUMMARY:
Study design to demonstrate the safety and performance of the Epitomee Device

DETAILED DESCRIPTION:
Prospective, single center, open-labeled single arm study. The subjects will be enrolled in one investigational site. Subjects meeting eligibility criteria will receive multiple capsule intakes, 1 capsule twice daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. 21 ≤ Age <65 years
2. 28 < BMI ≤ 40 kg/m2
3. Healthy subject
4. Normal blood count and chemistry
5. Subject is able and willing to give informed consent
6. Subject is able and willing to participate in the study and follow protocol procedures

Exclusion Criteria:

A. General health and medication

1. Any history or evidence of significant cardiac, renal, neurologic, pulmonary, gastrointestinal, hematologic abnormality, chronic hepatic disease or any other disease or symptom which in the judgment of the investigator would interfere with the study or confound the results
2. Symptomatic or unbalanced metabolic syndrome, or, symptomatic or unbalanced type 2 diabetes - such patients with minor symptoms may be allowed according to the PI discretion
3. Intake of chronic medication which may affect the GI or interrupt with the treatment, unless approved by the PI discretion
4. Taking thyroid hormone deficiency drugs (such as L-thyroxine)
5. Hemoglobin level under 11 gm/dl

   B. Weight loss history and status
6. Currently using pharmaceutical agents or food supplements for weight loss
7. History of weight reduction of more than 5% of total body weight in the past 6 months
8. Eating disorder such as anorexia, bulimia compulsory overeating or emotional eating*

   C. Specific GI history and status
9. History or evidence of any active liver disease. (abnormal liver functions: >1.5 times upper limit)
10. Subject with Inflammatory Bowel Disease (IBD)
11. Significant swallowing disorders
12. Less than 3 natural bowel movements per week
13. Past history of any gastrointestinal surgery (excluding uncomplicated appendectomy)
14. Malabsorption disorders

    D. General
15. History of food allergy according to PI decision
16. Female subjects who are breastfeeding or have a positive pregnancy test at screening or at any time during the study
17. History of alcohol or drug abuse within 6 months of screening
18. Mental disorders
19. Currently participating in an ongoing clinical study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-09-04 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Safety evaluation of the Device administration. | Baseline, 12 weeks
  Normal Gastroscopic examination as assessed by an independent safety committee.
the change in subjects' weight presented as percent total body loss (%TBL) | Baseline, 12 weeks
  Subjects loss of weight described as %TBL

CONTACTS AND LOCATIONS:
Overall Officials: Haim Shirin, MD, Principal Investigator — The Kamila Gonczarowski Institute of Gastroenterology Assaf Harofeh Medical Center,
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcomes measures will be made available
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available within six months of study completion